CLINICAL TRIAL: NCT04063995
Title: Effect of Repetitive Transcranial Magnetic Stimulation Over Contralesional Dorsal Premotor Cortex on Post Stroke Upper Limb Spasticity
Brief Title: Repetitive Transcranial Magnetic Stimulation in Post Stroke Upper Limb Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ilker şengül, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-KAE-0292
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Spasticity as Sequela of Stroke
Keywords: Spasticity; Stroke; Repetitive transcranial magnetic stimulation; Premotor cortex
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Excitatory repetitive transcranial magnetic stimulation group (Experimental): One session of repetitive transcranial magnetic stimulation (rTMS) treatment with 10 Hz frequency will be applied to the contralesional dorsal premotor cortex. Application will be performed with Neurosoft-Neuro MS / D device. 90% of the motor threshold will be used in the stimulation. Stimulation is planned for a total of 15 minutes and a total of 1500 beats in the form of a 5 seconds 10 Hz stimulation followed by a 25 seconds interval.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Inhibitory repetitive transcranial magnetic stimulation group (Experimental): One session of repetitive transcranial magnetic stimulation (rTMS) treatment at 1 Hz frequency will be applied to the contralesional dorsal premotor cortex. Application will be performed with Neurosoft-Neuro MS / D device. 90% of the motor threshold will be used in the stimulation. Stimulation is planned for a total of 25 minutes and a total of 1500 beats in the form of 1 Hz stimulation.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation group (Sham Comparator): Single session of sham application for a total of 25 minutes. Sham application will be performed by holding the probe of the device vertically to the vertex. The device will be operated at the lowest operating power of 1 to produce the same stimulation sounds like the active application. The device operating at this power is not likely to give any stimulation due to the probe being held upright.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive intervention that uses magnetic fields to stimulate nerve cells to improve the symptoms of a variety of disorders, including stroke-related motor impairment.

SUMMARY:
The reticulospinal pathway (RSP) is at the center of spasticity mechanism. The RSP indirectly synapses with motor neurons via interneurons in the ventromedial intermediate zone in both halves of the spinal cord, and directly synapses with motor neurons of proximal extremity muscles. The main motor cortex region controlling unilateral RSP is the premotor cortex. That is, a single limb is represented in both premotor cortices. This suggests theoretically that if the corticoreticular pathway controlling RSP is modulated by dorsal premotor cortex stimulation, there may be a change in the regulation of the intraspinal network regulating the stretch reflex. Therefore, the hypothesis in this study is that the application of repetitive transcranial magnetic stimulation (rTMS) over the contralesional dorsal premotor cortex in chronic stroke patients changes the severity of spasticity.

DETAILED DESCRIPTION:
Spasticity is a disorder characterized by increase in velocity-related muscle tone as a part of upper motor neuron syndrome. Although the mechanisms underlying stroke-related spasticity have not been fully understood, the current view is that spasticity is related to an imbalance between descending excitatory and inhibitory systems that regulate spinal stretch reflex and associated with abnormal intraspinal processes. The reticulospinal pathway (RSP) is at the center of this mechanism called cortical disinhibition. The dorsal RSP, which has an inhibitory effect on the spinal stretch reflex, originates from the medullary reticular formation and is under cortical control. In contrast to dorsal RSP, medial RSP which is not under the control of motor cortex originates from pontine reticular formation,and has an excitatory effect on spinal stretch reflex. The main motor cortex region controlling unilateral dorsal RSP is the premotor cortex. Unilateral RSP indirectly synapses with motor neurons via interneurons in the ventromedial intermediate zone in both halves of the spinal cord, and directly synapses with motor neurons of proximal extremity muscles. That is, a single limb is represented in both premotor cortices. This suggests theoretically that if the corticoreticular pathway controlling dorsal RSP is modulated by dorsal premotor cortex stimulation, there may be a change in the regulation of the intraspinal network regulating the stretch reflex. Furthermore, in stroke patients with severe motor impairment, the relationship between high cortical centers and the primary motor cortex is more in the form of facilitation rather than interhemispheric inhibition between the primary motor cortices. In other words, stimulation of one side premotor cortex may affect motor impairment and spasticity by affecting primary and high motor cortical centers of both hemispheres and both halves of the spinal cord. Therefore, the hypothesis in this study is that the application of repetitive transcranial magnetic stimulation (rTMS) over the contralesional dorsal premotor cortex in chronic stroke patients changes the severity of spasticity. Based on this hypothesis, our aim is to investigate the effect of rTMS over the contralesional dorsal premotor cortex on the severity of spasticity in patients with chronic stroke with moderate to severe upper extremity spasticity.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Stroke history ≥ 1 year
* Having a first stroke
* Grade 2 or 3 muscle tone according to the Modified Ashworth Scale (MAS) assessment in at least one of the elbow, wrist and finger flexors
* Signed consent to participate in the study

Exclusion Criteria:

* To have a clinical condition (metallic implant, cardiac pace, pregnancy, breastfeeding, claustrophobia, epilepsy, head trauma, cranial operation history) that will constitute a contraindication to transcranial magnetic stimulation
* Presence of malignancy
* Pregnancy or breastfeeding
* Non-stroke disease or lesion affecting the sensorimotor system
* Presence of pump/shunt
* Advanced cognitive impairment
* To have been rehabilitated in the last 3 months
* Botulinum toxin injection in the last 3 months
* Taking systemic antispastic drugs (Patients taking these drugs may be included in the study after a period of at least 3 times the half-life of the drug used if they agree to quit)
* Previously treated with TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Pre-intervention (baseline) and immediately after intervention (post-intervention), up to 45 minutes
  The modified Ashworth Scale is a scale that clinically evaluates the presence and severity of muscle tone increase. It is an ordinal scale that evaluates spasticity at six levels between 0 and 4 (0, 1, 1+, 2, 3, 4). The severity of spasticity increases as the score increases. Score 0 indicates no increase in muscle tone, while score 4 indicates that the affected part is rigid. Six levels between 0 and 5 (0, 1, 2, 3, 4, 5) will be used in statistical analysis. The score of 1+ will be treated as 2, 2 as 3, 3 as 4 and 4 as 5.

SECONDARY OUTCOMES:
F wave parameters | Pre-intervention (baseline) and immediately after intervention (post-intervention), up to 45 minutes
  F-wave is one of the late responses caused by antidromic stimulation of alpha motor neurons. It occurs following supramaximal electrical stimulation of peripheral motor nerves following M response. The F wave indicates the transmission from the stimulated point to the motor neuron and back to the recording electrode. Increased F wave frequency, increased F / M ratio and amplitude has been considered to indicate the increased motor neuron excitability.

CONTACTS AND LOCATIONS:
Overall Officials: İlker Şengül, M.D., Principal Investigator — İzmir Katip Çelebi University
Locations (1):
- İlker Şengül, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li S, Francisco GE. New insights into the pathophysiology of post-stroke spasticity. Front Hum Neurosci. 2015 Apr 10;9:192. doi: 10.3389/fnhum.2015.00192. eCollection 2015. PMID 25914638
- [Background] Burke D, Wissel J, Donnan GA. Pathophysiology of spasticity in stroke. Neurology. 2013 Jan 15;80(3 Suppl 2):S20-6. doi: 10.1212/WNL.0b013e31827624a7. PMID 23319482
- [Background] Lemon RN. Descending pathways in motor control. Annu Rev Neurosci. 2008;31:195-218. doi: 10.1146/annurev.neuro.31.060407.125547. PMID 18558853
- [Background] Baumer T, Bock F, Koch G, Lange R, Rothwell JC, Siebner HR, Munchau A. Magnetic stimulation of human premotor or motor cortex produces interhemispheric facilitation through distinct pathways. J Physiol. 2006 May 1;572(Pt 3):857-68. doi: 10.1113/jphysiol.2006.104901. PMID 16497712
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Wupuer S, Yamamoto T, Katayama Y, Motohiko H, Sekiguchi S, Matsumura Y, Kobayashi K, Obuchi T, Fukaya C. F-wave suppression induced by suprathreshold high-frequency repetitive trascranial magnetic stimulation in poststroke patients with increased spasticity. Neuromodulation. 2013 May-Jun;16(3):206-11; discussion 211. doi: 10.1111/j.1525-1403.2012.00520.x. Epub 2012 Oct 24. PMID 23094969
- [Derived] Sengul I, Askin A, Altun A, Tosun A. Anti-spastic effect of contralesional dorsal premotor cortex stimulation in stroke patients with moderate-to-severe spastic paresis: a randomized, controlled pilot trial. Acta Neurol Belg. 2023 Aug;123(4):1345-1354. doi: 10.1007/s13760-023-02212-2. Epub 2023 Feb 21. PMID 36809647